CLINICAL TRIAL: NCT02152111
Title: Effect of Hipoernergetic Diet Combined or Not With Coconut Flour on Overweight Women
Brief Title: Hipoenergetic Effect of Diet Associated or Not With the Consumption of Coconut Flour in Women With Overweight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Elizabeth de Paula Franco, Miss, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05155812.2.0000.5257
Record Dates: First submitted 2014-04-04; First posted 2014-06-02 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Obesity; Cardiovascular Risk Factor
Keywords: Obesity; Coconut flour; Diet quality; Cardiovascular risk factor
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement: Coconut flour (Experimental): Diet hipoernergetic plus 26g/day coconut flour during three months (12weeks).
  Interventions: Dietary Supplement: Coconut flour
- Nutritional Treatment (Active Comparator): All patients received an individualized diet plan and balanced. The diet was calculated to the nutritional status and the protein 15-20% of total energy value, lipids 25-30% of daily energy intake and carbohydrate 50-60% of total energy value
  Interventions: Behavioral: Diet

INTERVENTIONS:
Dietary Supplement: Coconut flour — Patients 9 months following treatment, starting at 3 months with diet hipoenergetica 3 months washout and sixth month diet hiponergetic more coconut flour.
  Arms: Dietary Supplement: Coconut flour
Behavioral: Diet — Patients were instructed to follow the dietary treatment for 6 months.
  Arms: Nutritional Treatment

SUMMARY:
This study aimed to evaluate the effect of weight loss with diet combined coconut flour consumption improvement weight loss and reduction in glucose, cholesterol in obese women.

DETAILED DESCRIPTION:
This is a clinical trial with two groups, one receiving hipoenergetic diet for 180 days and another group with hipoenergetic diet for 90 days, a washout period for another 90 days and another period for another 90 days diet meal plus hipoenergética coconut. In order to assess body mass, waist circumference and neck, assess the lipid profile, glucose and uric acid.

ELIGIBILITY:
Inclusion Criteria:

women > 20 years old BMI >25 Kg/m²

Exclusion Criteria:

Performing diets and / or making use of drugs for the reduction of body weight; Supplements of any kind; Pregnant and lactating women; In use of statins; With voluntary water restriction. -

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Anthropometry | 9 months
  To evaluate the effect to coconut flour in the improvement of weight, waist circumference and neck circumference in voluntary overweight and obesity

SECONDARY OUTCOMES:
Lipid profile | 9 months
  To evaluate the effect the coconut flour in lowering total cholesterol, triglycerides, LDL cholesterol and HDL cholesterol.
Quality of the diet | 9 months
  To evaluating the effect of treatment on the nutritional quality of the diet

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth P Franco, Nutricionist, Principal Investigator — Universidade Federal do Rio de Janeiro